CLINICAL TRIAL: NCT05146648
Title: Mechanism of Action for Effects From Automated Mechanical Peripheral Stimulation
Brief Title: Gondola Mechanism of Action
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: study withdrawn
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, David Putrino, Director of Rehabilitation Innovation for the Mount Sinai Health System; Associate Professor, Rehabilitation Medicine, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: STUDY-21-00837
Record Dates: First submitted 2021-11-23; First posted 2021-12-07 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2022-06

CONDITIONS: Chronic Stroke; Cerebral Palsy; Parkinson's Disease
Keywords: ambulation; sensory stimulation; mobility; neurological disorder
MeSH Terms: conditions — Cerebral Palsy; Parkinson Disease; Nervous System Diseases

STUDY DESIGN:
Intervention Model Description: Twenty adult individuals in the chronic phase of stroke, 20 people with cerebral palsy, 20 with Parkinson's Disease (intermediate stage) and 20 healthy volunteers will be randomized to receive sham or real AMPS intervention.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: A blinded evaluator will collect all the demographic (age, gender, time since injury, injury type), clinical and functional data of the participants. The investigator performing transcranial magnetic stimulation assessments will also be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Real AMPS (Active Comparator): AMPS therapy consists of mechanical stimulations applied to two specific points on both feet: the tip of the big toe (hallux) and the first metatarsal joint.
  Interventions: Device: Gondola AMPS
- Sham AMPS (Sham Comparator): AMPS therapy applied to two non-specific points on both feet.
  Interventions: Device: Gondola AMPS

INTERVENTIONS:
Device: Gondola AMPS — One treatment session lasts about two minutes and consists of the application of a mechanical pressure pulses on each of the points, one after the other, for a set duration (a few seconds), which is repeated several times in sequence.
  Other Names: Automated Mechanical Peripheral Stimulation

SUMMARY:
This study will investigate the clinical, functional and neurophysiological effects of automated mechanical peripheral stimulation (AMPS) via the Gondola device administered to patients with chronic stroke, cerebral palsy and Parkinson's Disease. Results will be collected using standardized outcome measures and a transcranial magnetic stimulation assessment protocol including electrical stimulation and electromyographic recording.

DETAILED DESCRIPTION:
The working hypothesis for this pre-post intervention study is that one session of AMPS will increase voluntary motor drive of the plantar-flexors (soleus) muscle. The primary outcome measure will be maximum voluntary contraction (MVC) of the soleus (measured by electromyography, EMG); the secondary outcome will be the MVC of the antagonist muscle, the tibialis anterior. Data will be collected before the first session compared to directly after. The same measures in sham-stimulated and healthy volunteers will serve as controls.

ELIGIBILITY:
Inclusion Criteria:

* age 18 to 80;
* chronic stroke lesion >6 months after a cerebrovascular accident OR diagnosis of cerebral palsy OR Parkinson's Disease;
* presence of some degree of motor function in the ankle flexor (Soleus motor power >1);
* able to ambulate 10 meters without physical assistance.

Exclusion Criteria:

* medically unstable condition;
* presence of other concurrent neurological illness;
* cognitive impairment (Montreal Cognitive Assessment score <23);
* presence of any potential TMS risk factor: damaged skin at the site of stimulation;
* presence of an electrically, magnetically or mechanically activated implant, an intracerebral vascular clip, or any other electrically sensitive support system;
* family history of medication-resistant epilepsy;
* past history of seizures or unexplained spells of loss of consciousness.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01-12 (Actual); Primary Completion 2023-01-12 (Actual); Study Completion 2023-01-12 (Actual)

PRIMARY OUTCOMES:
Change in Soleus MVC | pre and post-AMPS (baseline and 2 minutes)
  maximum voluntary contraction of the soleus muscle (measured by EMG)

SECONDARY OUTCOMES:
Change in Tibialis anterior MVC | pre and post-AMPS (baseline and 2 minutes)
  maximum voluntary contraction of tibialis anterior (measured by EMG)
Change in 10 meter walk test | pre and post-AMPS (baseline and 2 minutes)
  self-selected pace to determine gait speed

CONTACTS AND LOCATIONS:
Overall Officials: Gabriela Rozanski, Study Director — MOUNT SINAI HOSPITAL; David Putrino, PT, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Abilities Research Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Not applicable to study aims